CLINICAL TRIAL: NCT00240864
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel Group Study of Acetaminophen 1000 mg and Ibuprofen 400 mg in Postoperative Dental Pain
Brief Title: An Effectiveness and Safety Study of Acetaminophen 1000 mg and Ibuprofen 400 mg in Postoperative Dental Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002671
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Pain
Keywords: postoperative dental pain; acetaminophen; ibuprofen
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

ARMS (3):
- 001 (Experimental): acetaminophen
  Interventions: Drug: acetaminophen
- 002 (Experimental): ibuprofen
  Interventions: Drug: ibuprofen
- 003 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo
  Arms: 003
Drug: acetaminophen
  Arms: 001
Drug: ibuprofen
  Arms: 002

SUMMARY:
The purpose of this study is to determine the onset of pain relief from a single dose of acetaminophen and ibuprofen in subjects experiencing postoperative dental pain following the surgical extraction of at least three molars.

DETAILED DESCRIPTION:
The primary objective of this randomized, double-blind, placebo-controlled study is to determine the onset of analgesia following the administration of a single dose of 1000 mg of acetaminophen, 400 mg of ibuprofen or placebo in subjects experiencing acute postoperative dental pain secondary to the surgical extraction of at least three molars, with at least one being a partial or complete bony mandibular third molar impaction. After reporting moderate to severe pain following dental surgery, subjects record their baseline pain intensity and are treated with a single oral dose of acetaminophen, ibuprofen, or placebo. Subjects evaluate their pain intensity and pain relief relative to baseline at various timepoints up to 4 hours after taking study medication. Pain intensity is assessed using a five-point scale consisting of none (0), mild (1), moderate (2), moderately severe (3), and severe (4). Pain relief from baseline is evaluated on a five-point scale consisting of none (0), a little (1), some (2), a lot (3), and complete (4). At the end of the first hour of the observation period or at the time of taking supplemental analgesic medication (rescue treatment), whichever occurs first, subjects make an overall (global) assessment of the study medication, based on a five-point scale consisting of poor (0), fair (1), good (2), very good (3), or excellent (4). Subjects are required to remain at the study site for the duration of the four-hour observation period. The primary efficacy assessments are pain intensity differences from baseline and pain relief at each measurement time. Safety is assessed by monitoring adverse events occuring throughout the study. The primary hypotheses are that there is a difference between acetaminophen and placebo and between ibuprofen and placebo at some time point for the proportion of subjects reporting non-zero pain relief. The patients receive a single oral dose of one of the following three treatments: Two acetaminophen 500 mg caplets and two placebo ibuprofen capsules, two placebo acetaminophen caplets and two ibuprofen 200 mg capsules, or two placebo acetaminophen caplets and two placebo ibuprofen capsules.

ELIGIBILITY:
Inclusion Criteria:

* Indicates moderate to severe pain following the extraction of at least three molars (including at least one partial or complete bony mandibular third molar impaction)
* weighs at least 100 pounds and has a Body Mass Index (BMI) between 18 and 28
* not taking any medications for anxiety, depression or schizophrenia
* if female, not pregnant or breastfeeding

Exclusion Criteria:

* Used ibuprofen or acetaminophen within 12 hours preceding surgery or any other pain relievers or anti-inflammatory drugs within 24 hours preceding surgery
* have any gastrointestinal disease that would interfere with the absorption and excretion of study medications
* unable to swallow the study medication whole
* have any significant medical condition
* have a history of adverse reactions to acetaminophen, ibuprofen or any anesthetic agent used in the extraction

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Time at which the proportion of subjects indicating non-zero pain relief for each active treatment becomes statistically significantly superior to placebo.

SECONDARY OUTCOMES:
Pain intensity differences from baseline and pain relief at each measurement time; Area under the curve of pain relief scores at1 hour (TOTPAR1); Pain intensity differences at 1 hour (SPID1); Subjects' global assessment of pain relief at one hour

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: An Effectiveness and Safety Study of Acetaminophen 1000 mg and Ibuprofen 400 mg in Postoperative Dental Pain — http://download.veritasmedicine.com/PDF/CR002671_CSR.pdf